CLINICAL TRIAL: NCT05786326
Title: The Use of Multi Holes Fully Covered Metallic Stents Versus Uncovered and Partially Covered Metallic Stents in the Management of Malignant Biliary Obstruction: Randomized Parallel Clinical Trial.
Brief Title: Multihole Fully Covered Metallic Stents in the Management of Malignant Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, H Abdelkader, lecturer at tropical medicine department, faculty of medicine,Zagazig, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB #10426/1-3-2023
Record Dates: First submitted 2023-03-10; First posted 2023-03-27 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Malignant Biliary Obstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multiholes fully covered metaalic stents group (Experimental): Insertion of multiholes fully covered self-expandable metallic stents in the biliary tree through Endoscopic retrogrades cholangiopancreatography (ERCP)patients with malignant biliary obstruction.
  Interventions: Device: group 1
- parially covered metallic stents group (Active Comparator): Insertion of partially covered metallic stents in patients with malignant biliary obstruction.
  Interventions: Device: group 2
- unocoered metaalic stents group (Active Comparator): Insertion of uncovered metallic stents in patients with malignant biliary obstruction.
  Interventions: Device: group 3

INTERVENTIONS:
Device: group 1 — Insertion of fully covered self-expanding metallic stents with multi-holes (FCSEMS- MH) Biliary stent HANAROSTENT® CCC (M.I.Tech Co., Ltd, pyeongtaek, Korea) in a biliary tree through endoscopic retrograde cholangiopancreatography (ERCP) under general anesthesia by expertise in patients with malignant biliary obstruction
  Other Names: multiholes fully covered metallic stent
  Arms: multiholes fully covered metaalic stents group
Device: group 2 — Insertion of partially covered self-expanding metallic stents HANAROSTENT® Biliary (NCN) in the biliary tree through ERCP under general anesthesia by Expertise in patients with malignant biliary obstruction.
  Other Names: partially covered metallic stents
  Arms: parially covered metallic stents group
Device: group 3 — Insertion of uncovered self-expanding metallic stents (Biliary stent HANAROSTENT® NNN) (M.I.Tech Co., Ltd. Pyeongtaek, Korea) in a biliary tree through ERCP under general anesthesia by Expertise in patients with malignant biliary obstruction.
  Other Names: uncovered metallic stents
  Arms: unocoered metaalic stents group

SUMMARY:
multiholes fully covered metallic stents in the management of malignant biliary obstruction

DETAILED DESCRIPTION:
Malignant biliary obstruction is still a diagnostic and therapeutic challenge requiring a multidisciplinary approach. Most cases are inoperable at the time of diagnosis. Relieving the obstruction and normalizing the serum bilirubin level is usually the first step by biliary catheterization and stent placement.

Biliary stent placement has largely replaced surgical bypass for the palliation of malignant biliary obstruction. Rigid plastic stents, despite it is cheap and easily removed, but with limited duration of stent patency. Self-expandable metal stents (SEMS) have larger luminal diameters and provide longer patency time than rigid plastic stents. SEMS are composed of a variety of metals and can be uncovered, partially covered, or fully covered.

Uncovered stents are prone to obstruction by tumor growths; however, covered stents may block bile duct branches and are at risk of migration. A multihole self-expandable metallic stent was developed to prevent the obstruction of bile duct branches. In addition, the holes may prevent migration due to small ingrowths which reduce the tension of the membrane

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of malignant obstructive jaundice.
* Patient not eligible for surgery.
* Age above 18 years, any gender.

Exclusion criteria:

* Benign obstructive jaundice.
* Patient eligible for surgery.
* Failure to stent insertion.
* Patient not fit for ERCP and/or anaesthesia.
* Surgical and anatomical abnormalities interfere with endoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of multi holes fully covered metallic stents in management of malignant biliary obstruction | at 3 and 6 months follow up after stents ineration
  Detect the stent in his place. Patients clinically improved, and bilirubin decrease or reach normal values.

SECONDARY OUTCOMES:
Stent dysfunction (obstruction or migration) | after 3 and 6 months from stents insertion
  detect the stents dysfunction either obstruction or migration by clinical examination and abdominal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Magdy, profeesor, Study Director — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Sharkia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No